CLINICAL TRIAL: NCT06809816
Title: Efficacy of OsteoBor in Postmenopausal Osteoporosis: A Randomized, Double-Blinded, Placebo-Controlled Phase 2 Trial
Brief Title: Efficacy of OsteoBor in Postmenopausal Osteoporosis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tabriz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr. Saeid Safiri, Dr., Tabriz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 75397
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium pentaborate pentahydrate (Experimental): In this study, participants in the experimental group will receive 1000 mg of boron daily. OsteoBor will be administered orally, following the dosage recommendations provided by previous studies. Additionally, all participants will receive standard daily doses of 1200 mg of calcium and 800 IU of vitamin D3 supplements.
  Interventions: Drug: Sodium pentaborate pentahydrate
- Placebo (No Intervention): The placebo capsules used in the study will be visually identical to the OsteoBor capsules in terms of appearance and packaging. These capsules will be administered in the same way as the OsteoBor to maintain blinding and ensure that participants are unaware of their group allocation.

INTERVENTIONS:
Drug: Sodium pentaborate pentahydrate — Sodium pentaborate pentahydrate will be administered orally in capsule form, following the standard protocol outlined in the study design.
  Arms: Sodium pentaborate pentahydrate

SUMMARY:
This study aims to evaluate the impact of boron supplementation (OsteoBor) on bone health in postmenopausal women. The trial is a phase 2, randomised, double-blind, placebo-controlled study lasting one year

DETAILED DESCRIPTION:
Osteoporosis is a systemic condition that affects the skeleton, characterised by decreased bone density and the destruction of bone microstructure, resulting in increased fragility and a higher risk of fractures. It disproportionately affects postmenopausal women due to reduced estrogen production, which plays a crucial role in bone metabolism. The disease leads to significant health burdens, including fractures that decrease quality of life and increase healthcare costs. The World Health Organization (WHO) defines osteoporosis as a bone mineral density (BMD) score of T ≤ -2.5, and the prevalence of low BMD continues to rise globally, contributing to the increasing incidence of fractures.

This study evaluates OsteoBor, a boron-based supplement, for improving BMD and reducing fracture rates in postmenopausal women in Iran. Boron, a trace mineral, supports bone health by influencing calcium, magnesium, and vitamin D metabolism, and shows promise in reducing inflammation and enhancing antioxidant enzymes. Although animal studies have shown positive effects on bone mineralisation, human studies remain limited. This trial aims to explore the effectiveness of OsteoBor as a potential alternative to existing osteoporosis treatments, which face challenges like side effects and patient adherence.

ELIGIBILITY:
Inclusion Criteria:

Age Range: Postmenopausal women aged 45 to 85 years. Menopause status must be confirmed, with at least 1 year since the last menstrual period.

Bone Mineral Density (BMD): T-score at the lumbar spine, total hip, or femoral neck should be ≤ -2.5 but > -3.5.

General Health: Participants must be generally healthy with no significant chronic diseases that could affect bone health or the assessment of outcomes.

Compliance with OsteoBor: All participants must be willing to adhere to daily intake of OsteoBor or placebo, along with calcium (1200 mg) and vitamin D (800 IU) supplements throughout the study.

Informed Consent: Participants must sign written informed consent before enrolment and confirm their understanding of the study design, interventions, and potential risks.

-

Exclusion Criteria:

History of Fractures: A history of hip fractures or more than one clinical fracture in the spine. Any fractures other than hip fractures (except for fractures of fingers, toes, or the skull) within the past 24 months.

Other Bone Diseases: Presence of metabolic bone disorders other than osteoporosis, such as Paget's disease, osteomalacia, or hyperparathyroidism. Rheumatoid arthritis or other inflammatory joint diseases that could affect bone health.

Kidney-Liver Problems & Calcium Metabolism: Severe kidney failure, defined as serum creatinine levels above 1.6 mg/dL, or a history of kidney stones. Abnormalities in serum calcium levels, 25-hydroxy vitamin D, or parathyroid hormone (PTH) levels.

Prohibited Medications: Use of oral bisphosphonates in the past 6 months or long-term use (more than 6 months) at any time in the past. Any use of IV bisphosphonates, including zoledronate, in the year prior to the study. Use of denosumab, teriparatide, or any anabolic bone drug within the past 12 months. Use of systemic glucocorticoids (equivalent to more than 5 mg/day of prednisone) for over 2 weeks in the past 6 months. Use of active vitamin D, strontium ranelate, or other investigational bone health agents in the past 3 months.

Chronic Diseases: Diseases affecting bone metabolism or physical mobility, such as uncontrolled thyroid disease, uncontrolled diabetes, or severe gastrointestinal disorders that affect nutrient absorption. Any conditions that cause persistent tremors that might interfere with imaging or medication adherence.

Previous Participation in Other Studies: Recent participation in clinical trials involving investigational drugs or supplements for bone health within the past 12 months.

Alcohol and Drug Use: Heavy alcohol consumption (>2 drinks/day) or substance abuse that could affect study compliance and bone health.

Allergies and Sensitivities: Known allergies or sensitivities to boron supplements, calcium, vitamin D, or other components of the study drugs.

-

Ages: 45 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
The percentage change in areal bone mineral density (aBMD) | The measurements will be taken at baseline, 6 months, and 12 months.
  The change in areal bone mineral density (aBMD) at the lumbar spine will be evaluated over a 12-month period, comparing the baseline measurement to the final result. This will be assessed using dual-energy X-ray absorptiometry (DXA), a widely used and trusted technique for bone health evaluation. The lumbar spine is particularly important for assessing bone density, as it is a key area affected by osteoporosis, especially in postmenopausal women who are at higher risk of fractures due to changes in hormonal levels.

SECONDARY OUTCOMES:
The percentage change in aBMD at the total hip and femoral neck | At baseline, 6 months, and 12 months.
  It will be measured using dual-energy X-ray absorptiometry (DXA).
Serum Osteocalcin | At baseline, 6 months, and 12 months.
  Serum osteocalcin is a biomarker for bone formation, and its levels can help assess osteoporosis progression by reflecting the balance between bone resorption and formation. Decreased osteocalcin levels are associated with lower bone formation rates and higher fracture risk, especially in postmenopausal women
Bone-specific alkaline phosphatase | At baseline, 6 months, and 12 months.
  Bone-specific alkaline phosphatase (BSAP) is a marker of bone formation, primarily produced by osteoblasts, and is elevated in conditions like osteoporosis, reflecting increased bone turnover. Elevated BSAP levels can indicate active bone repair, while lower levels might suggest reduced bone formation, aiding in monitoring osteoporosis progression and treatment effectiveness

IPD SHARING:
Plan to Share IPD: Undecided